CLINICAL TRIAL: NCT00808925
Title: The Impact of Heat Acclimation on Pro- and Anti- Inflammatory Cytokine Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Yoram Epstein (Other Government)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor-Investigator, Prof. Yoram Epstein, Heller institue, Sheba Medical Center, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SHEBA-08-5524-YE-CTIL
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: "Exposure to Heat"
Keywords: acclimation; heat; cytokines; stress; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental)
  Interventions: Other: exposure to heat

INTERVENTIONS:
Other: exposure to heat — Dressed in shorts and tennis shoes the subjects will be exposed to exercise-heat stress for 12 consecutive days (excluding Saturday). Daily exposure will last 120 min, under the controlled environmental conditions of 40oC and 40% relative humidity. The exercise will consist of walking on a treadmill at a pace of 5km/h and 2% incline.
  Other Names: acclimation to heat

SUMMARY:
There is growing evidence to conclude that part of the cascade leading to heatstroke is related to an inflammatory reaction triggered by the heat stress. The reduced ability to sustain heat stress - "heat intolerance" is also attributed to over-expression of inflammatory cytokines. Acclimation to heat improves human sustainability to heat and is a leading protective factor against heat stroke. The investigators hypothesize that the lower stress encountered during the process of acclimation to heat will be reflected by an over-ride in the expression of anti-inflammatory over the pro-inflammatory cytokines. This, in turn will attenuate the pathological cascade leading to heat stroke.

ELIGIBILITY:
Inclusion Criteria:

* age:18-25
* medically screened (healthy)

Exclusion Criteria:

* BMI over 22 kg/m2
* systolic blood pressure over 120 mmHg
* any febrile illness during the last week preceding the study
* any skin disease
* diabetes
* any heart conditions.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Investigating the variability in the levels of different cytokine and the kinetics in cytokine levels during the process of acclimation to heat. | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Moran, PhD, Study Director — Institute of Military Physiology, IDF Medical Corps
Locations (1):
- Heller Institute of Medical Reachearch, Sheba Medical Center, Tel Litwinsky, Israel